CLINICAL TRIAL: NCT07218627
Title: A Randomised, Placebo-controlled, Double-blinded Phase 1b Study Investigating Safety, Tolerability, Pharmacokinetics and Effects on Biomarkers From Multiple Ascending Doses of NNC0537-1482 in Participants With Heart Failure
Brief Title: A Research Study on the Effects of NNC0537-1482 in Participants With Heart Failure
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6537-7866; U1111-1313-9985 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1A (Experimental): Participants will be administered once weekly dose level 1 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482
- Cohort 2A (Experimental): Participants will be administered once weekly dose level 2 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482
- Cohort 3A (Experimental): Participants will be administered once weekly dose level 3 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482
- Cohort 4A (Experimental): Participants will be administered once weekly dose level 4 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482
- Cohort 5A (Experimental): Participants will be administered once weekly dose level 5 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482
- Cohort B (Experimental): Participants will be administered a selected safe and tolerable dose level of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482
- Placebo (Placebo Comparator): Participants will be administered Placebo matched to NNC0537-1482 subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0537-1482 — NNC0537-1482 will be administered subcutaneously.
  Arms: Cohort 1A; Cohort 2A; Cohort 3A; Cohort 4A; Cohort 5A; Cohort B
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Placebo

SUMMARY:
The study is testing a new drug (NNC0537-1482) to potentially treat people with heart failure. The purpose of the study is to see if NNC0537-1482 is safe and how it works in the body. Participants will either get NNC0537-1482 or placebo (a "dummy drug" without any active ingredients) and which treatment they get is decided by chance. This study will last up to 64 days with an additional screening period up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or females of non-childbearing potential.
* Age 40-75 years (both inclusive) at the time of signing the informed consent.
* Body Mass Index (BMI) range 18.5 - less than (<) 40 kilogram per square meter (kg/m^2).
* Symptomatic heart failure (New York Heart Association class II-III).
* Stable standard of care medical therapy for heart failure with mildly reduced ejection fraction/heart failure with preserved ejection fraction (HFmrEF/HFpEF) defined by:
* No addition or removal of sodium-glucose cotransporter 2 inhibitors (SGLT2i), angiotensin-converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), beta-blockers (BBs,) calcium-channel blockers or aldosterone antagonists, and no substantial change in dosage (greater than or equal to (≥)100% increase/decrease) at least 4 weeks before screening.
* On a diuretic therapy at least 2 weeks before screening without substantial change in dosing (≥50% increase/decrease), and on a stable diuretic therapy at least 1 week before screening.
* On the stable doses (not in titration period) of standard medical therapy for other comorbidities
* No hospitalizations due to heart failure (HF) between screening (V1) and randomisation (V2) confirmed at randomisation.
* Left ventricle ejection fraction (LVEF) greater than (>) 40 percentage (%) documented by echocardiography at screening, or within 12 months prior to screening with no change in clinical status suggesting potential for deterioration in systolic function.

AND at least one of the following:

* N-terminal pro type-B natriuretic peptide (NT-proBNP) ≥125 picogram per milliliter (pg/mL) (for participants with sinus rhythm) or NT-proBNP ≥375 pg/mL (for participants with persistent/permanent atrial fibrillation) at screening, and ≥1 of the following (documented by echocardiography within 12 months prior to or at screening):
* Septal é <7 or lateral <10 or average E/é ≥10
* Pulmonary artery (PA) systolic pressure >35 millimeters of mercury (mmHg)
* Left atrium (LA) enlargement, (width ≥3.8 centimeter (cm) or length ≥5.0 cm or area ≥20.0 square centimeter (cm^2) or volume ≥55 milliliter (mL) or left atrial volume index (LAVI) ≥29 milliliter per square meter (mL/m^2)
* Left ventricular hypertrophy (LVH) with septal thickness or posterior wall thickness ≥1.2 cm.
* Hospitalization with a primary diagnosis of decompensated HF requiring intravenous loop diuretic treatment within previous 12 months, and ≥2 of the following (documented by echocardiography within 12 months prior to or at screening):
* Septal é <7 or lateral <10 or average E/é ≥10
* PA systolic pressure >35 mmHg
* LA enlargement, (width ≥3.8 cm or length ≥5.0 cm or area ≥20.0 cm^2 or volume ≥55 mL or LAVI ≥29 mL/m^2)
* LVH with septal thickness or posterior wall thickness ≥1.2 cm
* Ongoing use of diuretic therapy for ≥30 days before screening.
* Mean pulmonary capillary wedge pressure (PWP) ≥15 mmHg or left ventricular end-diastolic pressure (LVEDP) ≥15 mmHg documented during catheterization at rest or PA diastolic pressure measured by implantable monitor ≥15 mmHg or PWP or LVEDP ≥25 mmHg documented during catheterization at exercise.

Exclusion Criteria:

* Any prior echo measurement of LVEF less than or equal to (≤) 40%, under stable conditions, within the past 36 months.
* Previous participation in this study (defined as being randomised).
* Ongoing treatment with a neprilysin inhibitor (including angiotensin receptor/neprilysin inhibitor treatment), phosphodiesterase-5 (PDE5) inhibitors or soluble guanylate cyclase (sGC) stimulators.
* Acute coronary syndrome (ACS) (including myocardial infarction (MI)), stroke, transient ischemic attack (TIA), carotid surgery or angioplasty, cardiac surgery, other major cardiovascular surgery, or urgent percutaneous coronary intervention within the 3 months prior to screening.
* Current acute decompensated HF requiring augmented therapy.
* Hospitalisation within the last 90 days prior to screening with HF as the primary cause.
* Known or suspected hypersensitivity to study intervention(s) or related products.
* Probable alternative diagnoses that in the opinion of the investigator could account for the participant's HF symptoms (i.e., dyspnoea, fatigue) such as significant pulmonary disease (including primary pulmonary hypertension, severe chronic obstructive pulmonary disease), anaemia, hypothyroidism or obesity.
* Systolic blood pressure outside the range of 110-160 mmHg at screening or randomisation.
* Heart rate outside the range of 40-110 beats per minute (bpm) at screening or randomisation.
* Orthostatic hypotension (defined as a decrease in systolic blood pressure ≥20 mmHg or a decrease in diastolic blood pressure ≥10 mmHg from a supine position to standing after 3 minutes, at screening or randomisation).
* Atrioventricular-block II or III, QRS >120 milliseconds (ms), or QTcF interval >450 ms for men and >470 ms for women, or any other clinically significant abnormal electrocardiogram (ECG) results as judged by the investigator at screening or randomisation.
* Participant has pacemaker, or implantable cardioverter defibrillator (ICD), cardiac resynchronization therapy (CRT) or left ventricular assist device (LVAD).
* Life-threatening or uncontrolled dysrhythmia, including symptomatic or sustained ventricular tachycardia and atrial fibrillation or flutter with a resting ventricular rate >110 bpm at screening or at randomisation.
* Significant changes of prescription medicinal products (dose or frequency) or non-prescription drugs between screening and randomisation visits, per investigator's assessment.
* Blood donation, plasma donation or blood draw any of the circumstances below:
* 400 mL within the past 90 days prior to the day of screening
* 50 mL within the past 30 days prior to the day of screening.
* Coronary or carotid artery disease or valvular heart disease likely to require surgical or percutaneous intervention within the 3 months after screening.
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≥2 times upper limit of normal (ULN).
* Estimated glomerular filtration (eGFR) <20 milliliter per minute per 1.73 square meter according to 2021 CKD-EPI equation.
* History or presence of any other disease (i.e., including malignancies) with a life expectancy of <1 year at screening.
* Receiving insulin for the treatment of diabetes type 1 or diabetes type 2.
* Glycated haemoglobin (HbA1c) of > 8.0% as measured at screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAE) | From pre-dose on day 1 until completion of the end of study (day 64)
  Measured as number of events.

SECONDARY OUTCOMES:
Cmax,MD; the maximum plasma concentration of NNC0537-1482 after last dose | From pre-dose on day 22 until completion of the end of study (day 64)
  Measured in nanomoles per liter (nmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Richmond Pharmacology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com